CLINICAL TRIAL: NCT05971914
Title: Alveolar Cleft Hard- and Soft Tissue Reconstruction With an Autogenous Tooth Derived Particulate Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Nagy Krisztián, Associate Professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cleftgraft-Semmelweis
Record Dates: First submitted 2023-07-21; First posted 2023-08-02 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cleft Lip and Palate
Keywords: cleft lip and palate; split thickness flap; autogenous tooth bone graft
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: Eight patients aged 8-12 years exhibiting uni- or bilateral alveolar cleft defects and oronasal fistulas underwent supra-, subgingival scaling and received individual oral hygiene instructions prior to surgery at the Department of Periodontology, Semmelweis University, Budapest, Hungary. Surgeries will be performed at the I. Department of Paediatrics, Semmelweis University, Budapest, Hungary between January 2021 and November 2021. The study was approved by the Semmelweis University Regional and Institutional Committee of Science and Research Ethics (Approval Number SE TUKEB x/2020). Patients is treated in accordance with the World Medical Association Declaration of Helsinki (version 2008). Surgical interventions are undertaken with the understanding and written consent of each subject's caregiver
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autogenous tooth derived particulate graft and a novel split thickness papilla curtain flap (Experimental): Extracted deciduous teeth were prepared immediately after removal according to the manufacturer's instructions with the Bonmaker® device. Ready to use autogenous tooth bone graft (ATB) was mixed with fibrin glue in 3D planned and printed plastic cuvettes to obtain a sticky graft closely matching the shape and extent of the bony defect. The preshaped sticky ATB graft was inserted and compacted in the cleft defect. Subsequently, the tension-free split thickness flap was repositioned by shifting all buccal surgical papillae mesially to the adjacent or the second adjacent interproximal space, depending on the horizontal extent of the cleft.
  Interventions: Procedure: Autogenous tooth derived particulate graft and a novel split thickness papilla curtain flap

INTERVENTIONS:
Procedure: Autogenous tooth derived particulate graft and a novel split thickness papilla curtain flap — Extracted deciduous teeth were prepared immediately after removal according to the manufacturer's instructions with the Bonmaker® device. Ready to use autogenous tooth bone graft (ATB) was mixed with fibrin glue in 3D planned and printed plastic cuvettes to obtain a sticky graft closely matching the shape and extent of the bony defect. The preshaped sticky ATB graft was inserted and compacted in the cleft defect. Subsequently, the tension-free split thickness flap was repositioned by shifting all buccal surgical papillae mesially to the adjacent or the second adjacent interproximal space, depending on the horizontal extent of the cleft.

SUMMARY:
The present study aims at clinical and radiographic evaluation of the safety and efficacy of Bonmaker ATB powder combined with a novel split thickness papilla curtain flap in the treatment of alveolar cleft defects.

ELIGIBILITY:
Inclusion Criteria:

* children with alveolar cleft
* patient presented at least three deciduous teeth scheduled for extraction.

Exclusion Criteria:

* major relevant clinical diseases,
* systemic use of steroids,
* current or previous intravenous bisphosphonate treatment,
* acute infection at the operation site.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Radiological volumetric measurements | 6 months
  Volumetric measurements will be conducted after the healing period. On prealigned pre- and postoperative CBCT cross-sections, linear measurements and volumetric measurements will be taken parallel to a reference base to determine the width of the surgical area.

SECONDARY OUTCOMES:
soft tissue healing | during the 6 months postoperatively
  Healing of soft tissues was recorded via photo documentation.
complications | 1, 14, 30 days and 3 and 6 months after surgeries.
  Every complication will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No